CLINICAL TRIAL: NCT05313880
Title: Digital Tools in Heart Failure - a Survey of Patient Usage (DIGITAL-HF)
Brief Title: DIGITAL-HF - Digital Tools in Heart Failure - a Survey of Patient Usage (DIGITAL-HF)
Acronym: DIGITAL-HF
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 307636
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: Digital technology; Digital literacy; Patient activation measures
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Digital tool Survey: Sequential patients from the 4 heart failure clinics at our institution will be offered to take part in the study.

SUMMARY:
Heart failure is a chronic health condition associated with significant symptoms, an increased need of support from the NHS, and typically is associated with a reduction in life expectancy. The covid pandemic has made it more difficult for the NHS to deliver high quality care to the 1 million patients living with heart failure in the UK. NHS England plans that digitalisation of services will help, increasing efficiency and improving ability of patients to self-care and manage their conditions. "Digitalisation" includes the use of digital tools for health, such as Apps and online resources & support. But the typical heart failure patient does not receive a diagnosis of heart failure until their 70s or 80s, creating a significant risk of digital exclusion. The heart failure failure community doesn't have any information about which tools (if any) heart failure patients are using, or why.

Patients who attend the heart failure clinic at the Royal Brompton, either face-to-face or virtually, will be eligible for our study. They will be provided an information sheet and asked for informed consent. The study consists of 4 short questionnaires (30 questions total) which only takes between 10-15 minutes to complete, this consists of 3 previously validated questionnaires and one bespoke questionnaire related to their digital tool use.

The investigators aim to recruit 130 patients to help us better understand how many NHS patients with heart failure access digital tools, which ones are most often used, and how this relates to their health literacy, digital health literacy and overall attitude to their health condition and management. The investigators aim to describe different digital subgroups of patients and will use this information to help inform local and national policy around digital support for people living with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who attends one of the heart failure clinics at the Royal Brompton hospital with a diagnosis of heart failure will be considered for the study.

Exclusion Criteria:

* Unable to complete a questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a study of outpatients with a diagnosis of heart failure, regardless of ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Proportions of digital tool use | 6 months
  Proportions of study participants using a variety of digital tools to access information about heart failure including websites, mobile applications and social media. The frequency of use and reasons for use.
Correlation of digital tool use with demographics | 6 months
  The correlation between digital tool use and several patient demographics including age in years, gender, highest educational level in grade, estimated income in British pounds and ethnic group.
Correlation of digital tool use with measures of patients' heart failure | 6 months
  The correlation between digital tool use and left ventricular ejection fraction in percentage, time from diagnosis of heart failure in months, New York Heart Association classification of heart failure (NYHA) and number of comorbidities.
Correlation of digital tool use with validated questionnaires | 6 months
  The correlation between digital tool use and health literacy (as measured by the validated AAHLS questionnaire - All aspects of health literacy scale).
  The correlation between digital tool use and digital health literacy (as measured by the validated eHEALS questionnaire).
  The correlation between digital tool use and patient activation (as measured by the validated PAM®). Patient activation is the knowledge, skills and confidence to manage one's health and healthcare.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Cowie, Principal Investigator — Royal Brompton hospital, part of Guys and St Thomas' hospital
Locations (3):
- United Kingdom (3):
  - Royal Brompton Hospital, London
  - Guy's and St Thomas' foundation NHS trust, London
  - King's college NHS foundation trust, London

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF